CLINICAL TRIAL: NCT03880656
Title: Autologous Bone Marrow Mononuclear Cell Administration for Lower Extremity Compartment Syndrome Injury
Brief Title: BM-MNCs for Lower Extremity Compartment Syndrome Injury
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kenton W. Gregory, Director, Oregon Center for Regenerative Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018011
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Compartment Syndrome Traumatic Lower Extremity
Keywords: mononuclear cells

STUDY DESIGN:
Intervention Model Description: This is a two-stage, randomized, unblinded, multicenter (two sites), controlled phase 1 clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Autologous BM-MNCs High Dose (Experimental): Administration of autologous bone marrow mononuclear cells at High dose (700,000 cells/cc of tissue)
  Interventions: Biological: Intramuscular administration of autologous BM-MNCs
- Observational Control (No Intervention): Standard of care provided for subjects that have undergone a fasciotomy following a diagnosis of compartment syndrome. No autologous bone marrow mononuclear cells will be administered.
- Autologous BM-MNCs Low Dose (Experimental): Administration of autologous bone marrow mononuclear cells at a Low dose (350,000 cells/cc of tissue)
  Interventions: Biological: Intramuscular administration of autologous BM-MNCs

INTERVENTIONS:
Biological: Intramuscular administration of autologous BM-MNCs — Intramuscular administration of autologous BM-MNCs at either a low or high cell dose.
  Arms: Autologous BM-MNCs High Dose; Autologous BM-MNCs Low Dose

SUMMARY:
This is a phase 1 study to assess safety and tolerability of intramuscular administration of two different doses of autologous bone marrow mononuclear cells (BM-MNCs) for treatment of lower extremity injury complicated by compartment syndrome injury.

DETAILED DESCRIPTION:
The primary objectives are to assess safety and tolerability of a high and low dose of autologous bone marrow mononuclear cells. Secondary objectives include evaluation of potential responses of the BM-MNC therapy.

This is a two-stage, randomized, unblinded, multicenter (two sites), controlled phase 1 clinical trial to evaluate the safety of two different doses of intramuscular injections of autologous bone marrow mononuclear cells, commonly known as a type of stem cell. Acute compartment syndrome injury is a mixed soft tissue injury due to a trauma that causes edema leading to excessive pressure in the muscle compartment. This type of injury frequently results in permanent reduction in function and disability.

A total of 18 participants that have undergone a fasciotomy for treatment of a lower leg compartment syndrome will be enrolled with 6 assigned to the control (observational) group, 6 to the low cell-dose group and 6 to the high cell-dose group. The treatment arm will receive a single dose (high or low) of autologous BM-MNCs 5 - 9 days post injury and fasciotomy and a minimum of 3 months of standard of care physical rehabilitation. An observational control arm will not receive cells post fasciotomy but will undergo a standard of care course of physical therapy and will be followed for comparison to assess early safety signals and potential benefit.

ELIGIBILITY:
Inclusion Criteria:

* Females and males 18 - 70 years old
* Has single or multiple compartment syndrome of the lower leg that includes the anterior tibial compartment
* Trauma patients with lower extremity CS requiring fasciotomy that can be treated with autologous BM-MNC therapy on day 5-9 post-fasciotomy
* Ability to sign an informed patient consent form
* Access and willingness to complete a standard of care course of rehabilitation therapy and 24 months follow-up evaluations
* Ability to close the fasciotomy wound per physician assessment
* Anterior compartment muscle volume between 100 - 280 cc as determined by MRI/CT
* Within the institutions' clinical reference ranges for HbA1C
* Negative HIV test

  · - Non-fracture, closed fracture or compound fracture type I (wound less than 1cm & compound from within out) (Gustilo-Anderson classification)
* Female subjects must be of non-childbearing potential or must be using adequate contraception
* If female subject is of childbearing potential, subject must have a negative pregnancy test at screening
* Willing and able to adhere to the study schedule

Exclusion Criteria:

* Prior compartment syndrome of same limb;
* Active malignancy or has undergone treatment for a malignancy in the preceding 5 years as indicated in past medical history or self-report if medical records do not accompany subject or are unable to be collected (basal cell carcinoma non-exclusionary);
* HIV positive as indicated by past medical history, self-report, or positive HIV test;
* Diagnosis of Type 1 or Type 2 diabetes with elevated HbA1C consistent with diabetes;(controlled diabetes acceptable, diabetes medication for other diagnosis acceptable)
* Diagnosis of chronic lower extremity vascular disease as diagnosed by current physician diagnosis, indicated in past medical history, or self-report if medical records do not accompany subject or are unable to be collected;
* Patients unable to sign an informed patient consent;
* Anticipated amputation of involved limb;
* Neurological conditions (i.e. spinal cord injury or traumatic brain injury) that may prevent full participation in CS rehabilitation or potentially confound study outcome measures (i.e. balance and gait) per physician discretion
* Current systemic infection;
* Local infection of the involved muscle group;
* Use of ventilator that would preclude rehabilitation protocols;
* Lack of access or unwillingness to complete standard of care course of physical therapy rehabilitation;
* Life expectancy 12 months or less;
* Bone marrow disorders (i.e. leukemia, aplastic anemia, lymphoma) ;
* Inability to close the fasciotomy wound or lower extremity burns that may affect wound closure
* Extensive tissue loss due to debridement resulting in insufficient residual tissue for stem cell administration and subsequent engraftment
* Lower extremity compound fracture type II or III (Gustilo-Anderson classification);
* Anterior tibialis muscle volume less than 100 cc or greater than 280 cc as determined by MRI/CT;
* Evidence of any past or present clinically significant medical condition that would impair wound healing
* History or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study as determined by the investigator or the investigator's designee;
* Any reason, considered by the principal investigator or designee, to preclude subject enrollment in the study that might represent a threat to the subject's health or safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety as determined by incidence of combined adverse events related to study agent intervention | Enrollment through 24 months
  Local and systemic reactions, serious adverse events and unexpected serious adverse events.
Efficacy as determined by muscle strength | 6 weeks, 3 months, 6 months, and 12 months
  Change in muscle strength compared to baseline and contralateral leg as measured by manual muscle testing and Biodex.

SECONDARY OUTCOMES:
Safety as determined by evidence of tumor formation | Baseline through 12 months
  Magnetic resonance imaging (MRI) and/or computed tomography (CT)
Efficacy as determined by muscle regeneration | Baseline through 12 months
  Magnetic resonance imaging (MRI) and/or computed tomography (CT) to measure muscle volume
Nerve conduction | Baseline and 6 months
  Nerve conduction velocity test
Wound healing | Baseline through 12 months
  Number of days until wound closure at the site of fasciotomy of the anterior compartment.
Lower extremity sensation | Baseline through 12 months
  Sensation as measured by Semmes Weinstein Monofilament.
Ankle range of motion | Baseline through 12 months
  Range of Motion (ROM): active and passive dorsi/plantar flexion ROM assessed using a goniometer.
Gait analysis | Week 6 through 12 months
  Change in gait kinematics: gait will be recorded using a Tekscan Pressure Mapping system where each sequential footstep is recorded along with synchronized video.
Gait endurance | Week 6 through 12 months
  Gait endurance measured using the 6-Minute Walk Test.
Gait speed | Week 6 through 12 months
  Gait speed measured using the 10 Meter Walk Test.
Balance | Week 6 through 12 months
  Balance assessed by single limb stance time.
Questionnaire - Pain | Baseline through 24 months
  Pain measured using the Numeric Pain Rating Scale (NPRS). The participant is asked to make three pain ratings (0 to 10; 0 - no pain, 10 - worst pain), corresponding to current, best and worst pain experienced over the past 24 hours. The average of the 3 ratings is used to represent the patient's level of pain over the previous 24 hours.
Questionnaire - Function | Baseline through 24 months
  Lower extremity function assessed using the Lower Extremity Functional Scale (LEFS). Total score (0 to 80; higher score = better outcome) is reported as a sum of 20 responses regarding functional activities (0 - extreme difficulty or unable to perform, 4 - no difficulty).
Questionnaire - Physical Activity | Baseline through 24 months
  Physical activity measured by the international physical activity questionnaire (IPAQ). Scores are reported as categorical (low, moderate, high) and/or continuous (metabolic equivalent minutes per week).

CONTACTS AND LOCATIONS:
Overall Officials: Kenton W Gregory, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No